CLINICAL TRIAL: NCT06006234
Title: The Status and Influencing Factors Analysis of Anxiety and Depression Among Residents of Elderly Care Institutions in Zhejiang Province
Brief Title: Analysis of Anxiety and Depression Among Elderly People
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: I2023616
Record Dates: First submitted 2023-07-31; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-07

CONDITIONS: Depression, Anxiety; Age Problem
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- residents of elderly care institutions: residents of elderly care institutions
  Interventions: Other: questionnaire survey

INTERVENTIONS:
Other: questionnaire survey — questionnaire survey

SUMMARY:
This study is a single-center, cross-sectional, and survey study. Through questionnaire surveys, information about the anxiety and depression status of residents of elderly care institutions in Zhejiang Province is collected. Through multi-factor analysis, the relevant influencing factors that affect their psychological status are clarified. The happy old age society provides reference opinions.

DETAILED DESCRIPTION:
China is one of the countries with the fastest aging population in the world. With the rapid aging of the population, there is an urgent need to build cities and communities into age-friendly cities and communities that facilitate the lives of the elderly and continue to make meaningful contributions to society. Various parts of our country are also actively exploring and constructing elderly care models with local characteristics, and an aging social environment of "respecting, loving and enjoying the elderly" is gradually being built.

However, due to the gradual decline of various organ capabilities with age, the elderly population has a higher risk of disease than other age groups. At the same time, due to limited income, the economic burden of the elderly population increases sharply after illness, and the quality of life is also affected to a certain extent. . According to a number of studies in recent years, the prevalence of depression in the elderly population is 26.0%, and the prevalence of anxiety disorders is 25.0%, which seriously affects the quality of life of elderly patients. With the progress of aging in our country, elderly care institutions are becoming more and more popular, and the elderly living in elderly care institutions often lack family companionship and social attention, and more psychological problems of the elderly may appear and be ignored.

Chronic diseases, different lifestyles, and pension forms are closely related to the mental health of the elderly, and at the same time affect the quality of life and social relationships of the elderly, thereby affecting disease recovery and survival. Therefore, it is particularly important to clarify the status quo of mental health and the prevalence of anxiety and depression among residents of nursing homes. At the same time, clarifying the relevant influencing factors will help researchers and related institutions to designate intervention measures, which has positive significance for social pensions.

This project intends to study the status quo of anxiety and depression among residents of nursing homes in Zhejiang Province, and at the same time analyze the factors related to depression and anxiety in the elderly, clarify the degree of effect of different factors, and provide guidance for nursing homes to improve the mental health of residents and improve life treatment. It is more in line with the pension model of an aging society.

ELIGIBILITY:
Inclusion Criteria:

* 1) ≥65 years old, lived in a nursing home for ≥1 year.
* 2) Not limited to men and women.

Exclusion Criteria:

* Those who cannot cooperate to complete the questionnaire, such as senile dementia, those who cannot express themselves after traumatic brain injury

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: residents of elderly care institutions in Zhejiang Province over 1 year
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
anxiety | 1 month
  anxiety score
depression | 1 month
  depression score

CONTACTS AND LOCATIONS:
Locations (1):
- Second affiliated hospital, school of medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No